CLINICAL TRIAL: NCT01444365
Title: A Phase 2, Randomized Withdrawal Study of the Analgesic Efficacy and Safety of ABT-652 as an Add On Therapy in Subjects With Osteoarthritis of the Knee Experiencing Partial Benefit of a Nonsteroidal Anti-Inflammatory Drug
Brief Title: A Study of ABT-652 in Combination With a Nonsteroidal Anti-Inflammatory Drug (NSAID) in Adults With Osteoarthritis Pain of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M13-237
Record Dates: First submitted 2011-09-28; First posted 2011-09-30 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABT-652 NSAID (Experimental): ABT-652 capsules -2 ABT-652 capsules twice daily (add-on) NSAID - as prescribed
  Interventions: Drug: ABT-652 NSAID
- Placebo NSAID (Placebo Comparator): Placebo - 2 placebo capsules twice daily NSAID - as prescribed
  Interventions: Drug: Placebo NSAID

INTERVENTIONS:
Drug: ABT-652 NSAID — ABT-652 capsules - 2 ABT-652 capsules twice daily (add-on) NSAID- as prescribed
  Arms: ABT-652 NSAID
Drug: Placebo NSAID — Placebo - 2 placebo capsules twice daily NSAID- as prescribed
  Arms: Placebo NSAID

SUMMARY:
To evaluate the safety and efficacy of ABT-652 in combination with a Non-steroidal Anti-inflammatory Drug (NSAID) compared to NSAID alone in adults with osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
This is a randomized withdrawal design study, containing a 4 week open-label period followed by a 6 week double-blind period. The total treatment period will be 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* History of osteoarthritis (OA) of the knee joint and meeting American College of Rheumatology (ACR) Clinical and Radiographic criteria,
* Currently taking nonsteroidal anti-inflammatory drugs (NSAIDs) and still experiencing pain as per the protocol requirements.
* Willing to washout of analgesics and to follow treatment plan, visit schedules and study procedures.

Exclusion Criteria:

* Diagnosis of rheumatoid arthritis, autoimmune disorder, arthritis other than osteoarthritis involving the study joint, or other painful syndrome that could interfere with the assessment of pain at the study joint
* Any cardiac, respiratory, neurological, psychiatric disorder or any other medical condition or illness that is not well controlled with treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Subject's Assessment of Arthritis Pain Intensity | 6 weeks
  Subject reported 24-hour average pain score measured by Visual Analogue Scale

SECONDARY OUTCOMES:
Western Ontario and McMaster (WOMAC™ ) Osteoarthritis Index | 6 weeks
  Self administered, patient-centered, health status questionnaire
Subject's Global Assessment of Arthritis Status | 6 weeks
  Subject reported pain intensity measured by Visual Analog Scale
Cognitive Functioning in Patients with Chronic Pain | 6 weeks
  Subject reported assessment of cognitive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Nothaft, MD, Study Director — AbbVie
Locations (31):
- United States (31):
  - Site Reference ID/Investigator# 61226, Phoenix, Arizona
  - Site Reference ID/Investigator# 61221, Phoenix, Arizona
  - Site Reference ID/Investigator# 61241, Tucson, Arizona
  - Site Reference ID/Investigator# 61257, Anaheim, California
  - Site Reference ID/Investigator# 61246, Fresno, California
  - Site Reference ID/Investigator# 61242, La Mesa, California
  - Site Reference ID/Investigator# 61204, Long Beach, California
  - Site Reference ID/Investigator# 61258, North Hollywood, California
  - Site Reference ID/Investigator# 61265, Milford, Connecticut
  - Site Reference ID/Investigator# 61234, DeLand, Florida
  - Site Reference ID/Investigator# 61213, Ocala, Florida
  - Site Reference ID/Investigator# 61211, Oldsmar, Florida
  - Site Reference ID/Investigator# 61217, Orlando, Florida
  - Site Reference ID/Investigator# 61231, Plantation, Florida
  - Site Reference ID/Investigator# 61245, Tampa, Florida
  - Site Reference ID/Investigator# 61263, Marietta, Georgia
  - Site Reference ID/Investigator# 61210, Brockton, Massachusetts
  - Site Reference ID/Investigator# 61260, Watertown, Massachusetts
  - Site Reference ID/Investigator# 61244, Florissant, Missouri
  - Site Reference ID/Investigator# 61266, St Louis, Missouri
  - Site Reference ID/Investigator# 61206, Omaha, Nebraska
  - Site Reference ID/Investigator# 61223, Salisbury, North Carolina
  - Site Reference ID/Investigator# 61273, Cincinnati, Ohio
  - Site Reference ID/Investigator# 61228, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 61264, Portland, Oregon
  - Site Reference ID/Investigator# 61238, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 61205, Beaumont, Texas
  - Site Reference ID/Investigator# 61218, Bryan, Texas
  - Site Reference ID/Investigator# 61235, San Antonio, Texas
  - Site Reference ID/Investigator# 61232, Draper, Utah
  - Site Reference ID/Investigator# 61269, Franklin, Wisconsin